CLINICAL TRIAL: NCT03377660
Title: The Effect of Clinical Treatment for Unintentional Weight Loss on Food Reward and Appetitive Behaviour in Patients Who Have Lost >10% of Their Body Weight After Undergoing Curative Surgery for Oesophageal Cancer
Brief Title: Resection of the Esophagus and Subsequent Weight Loss
Acronym: REWARD
Status: Terminated | Type: Observational
Why Stopped: Funding stopped.
Sponsor: Imperial College London (Other)
Collaborators: University College Dublin (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Carel Le Roux, Professor of experimental pathology, Reader in investigative science, Imperial College London
Other Study IDs: CRFSJ0148
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Cancer; Weight Gain; Eating Behavior; Food Reward
Keywords: Esophagectomy; Unintentional weight loss; Gut hormones
MeSH Terms: conditions — Esophageal Neoplasms; Weight Gain; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sandostatin: This cohort will be the group who are undergoing routine clinical treatment with a long-acting somatostatin analogue to minimise abnormal gut hormone signalling, and thus reduce early satiety.
  Interventions: Other: Clinical treatment
- Mirtazapine: This cohort will be the group who are undergoing routine clinical treatment with a tetracyclic antidepressant to stimulate appetite.
  Interventions: Other: Clinical treatment

INTERVENTIONS:
Other: Clinical treatment — Patients undergo clinical treatment as indicated, they are studied before and after.

SUMMARY:
The investigators aim to ascertain how food reward signals and eating behaviour relates to the gut-brain pathway in weight-losing patients after curative surgery for oesophageal cancer, and how this pathway responds to clinical treatment for this unintentional weight loss. The primary outcomes are the blood oxygen level dependent (BOLD) signal on functional MRI (fMRI), and the breakpoint during the progressive ratio task (PRT - a measure of eating behaviour), how these differ in response to multiple clinical treatment options, as well as how they relate to weight gain while on treatment.

DETAILED DESCRIPTION:
The incidence of cancer of the oesophagus (food pipe) is increasing. Improvements in treatment strategies have resulted in more people who remain free from cancer recurrence in the long term following treatment.

Surgery is the cornerstone of treatment for patients with oesophageal cancer, but while surgical removal of the tumour (oesophagectomy) may offer the best chance of cure, these are major operations associated with specific long term complications. Poor appetite, weight loss and nutritional impairment are common problems among patients who attain long-term cancer remission and cure after surgery.

A new clinic has been established to treat patients who are in remission but who have lost more than 10% of their body weight secondary to the effects of the surgery and struggling to regain weight. These patients will be treated as per standard of care with medications to aid weight gain.

The investigators are interested to conduct research into how the reward value of food changes during the clinical treatment pathway. The hypothesis is that there will be an increased reward response to food after medication use, the magnitude of which will correlate with weight gain. To assess this, patients who are already part of this clinic will be approached to have fMRI that can demonstrate changes in brain reward centres as well as a Progressive Ratio Task, which is a direct measure of appetitive behaviour. Changes in brain reward centre responses and appetitive behaviour will be correlated with changes in weight after pharmacotherapy. This may further inform future clinical protocols to provide improved precision medicine.

ELIGIBILITY:
Inclusion Criteria:

1. History of esophagectomy with gastric conduit reconstruction
2. Recurrence-free at least 12 months post-operatively
3. Weight loss ≥10% from premorbid weight, or requiring ongoing caloric supplementation
4. Due to undergo clinical treatment for weight loss with Sandostatin or Mirtazapine

Exclusion Criteria:

1. Pregnancy, breastfeeding
2. Significant and persistent chemoradiotherapy and/or surgical complication
3. Other active malignancy
4. Exocrine pancreatic insufficiency detected using fecal elastase
5. Uncontrolled diabetes mellitus
6. Significant psychiatric disorder or cognitive decline or communication impairment limiting capacity to provide informed consent
7. Severe dysphagia
8. Other disease or medication which may impact gut hormone physiology
9. History of significant food allergy, certain dietary restrictions
10. Any definite contraindication to somatostatin analogue administration
11. Claustrophobia, or any absolute contraindication to MRI scanning
12. Metallic implants, precluding fMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of post-esophagectomy patients at least 1 year after curative surgery, but struggling with unintentional weight loss of at least 10% baseline body weight, and thus candidates for clinical treatment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in BOLD signal | Before and after 4 weeks of clinical treatment
  Measure of food reward on fMRI
Change in breakpoint at PRT | Before and after 4 weeks of clinical treatment
  Measure of drive to eat

SECONDARY OUTCOMES:
Correlation of weight change during treatment with BOLD signal changes | Before and after 4 weeks of clinical treatment
  Relationship of food reward changes to weight gain
Correlation of weight change during treatment with PRT breakpoint changes | Before and after 4 weeks of clinical treatment
  Relationship of eating behaviour changes to weight gain

CONTACTS AND LOCATIONS:
Locations (1):
- Conway Institute, UCD, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No